CLINICAL TRIAL: NCT05932628
Title: Outcome and Prognosis of Supported Self-management in Thumb Base Osteoarthritis: A Prospective Cohort Study
Brief Title: Thumb Osteoarthritis Prognosis for Supported Self-managment
Acronym: TOPS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2021/042
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis Thumb
Keywords: Education; Exercise; Splint; Prognosis; Experience; Quality of care; Mixed Methods
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study will observe participants who receive a supported self management approach for thumb base osteoarthritis but it is not an interventional study. — Participants will receive an occupational or physiotherapist led supported self-management programme, which equates to normal NHS care, having been adopted by the sites involved. This involves education, progressive exercises and hand splints if required. The educational materials used, and a minimum number of appointments will be consistent across the study sites. Additional treatments for coexisting conditions will be provided, additional stepped care for thumb base osteoarthritis will also be recorded.

SUMMARY:
Background Thumb base osteoarthritis (OA) is common in adults 40 years and over. It affects a person's ability to work, be independent and care for others. Sufferers complain of severe pain and difficulty in completing everyday tasks. The main treatment for the condition is advice on how a person can manage their condition (self-management), reduce their pain, strengthen their hands with exercises and practical tips on tackling painful tasks, sometimes providing a hand splint for support. The treatment is provided by occupational and physiotherapists. We know that this treatment helps suffers in the short term (up to three months). But the research was done in people with few other health problems and while self-management support helps provide pain relief for most people, there are some people who don't benefit. The aim of this research is to see how pain and other hand problems change over a period of six months after the start of treatment, to understand people's experience of care, and examine why some people improve, and some do not.

Research Plan In patients receiving treatment for thumb base OA at four NHS sites, who are willing to take part, this research will: -

1. Record changes in symptoms and quality of life at three and six months from when treatment began in a postal questionnaire/survey.
2. Discuss the experience of care and people's beliefs about what makes treatment a success by interviewing a small group of patients.
3. Analyse patient characteristics, to see if it is possible to determine how they will respond to treatment.
4. Develop recommendations for improving care.

DETAILED DESCRIPTION:
Background

Thumb base osteoarthritis occurs in 21-45% of the adult population over 40 and can cause severe pain and difficulty with essential everyday hand use. Guidelines recommend that those seeking care should receive education and exercises (supported self-management), and, if needed, splints. However, these guidelines are based on research reporting outcomes at three months or less, often excluding those with other hand conditions and co-morbidities. In these studies, self-management was found to provide pain relief for about half of study participants, with the remaining individuals not benefiting significantly in terms of pain at three months. Furthermore, there is no research on the patient's experience of care.

The aim of this study is to investigate, using a mixed methods approach the outcomes, prognosis, and experiences of care in patients receiving usual National Health Service (NHS) care which consists of a supported self-management programme, and to generate recommendations for optimising care for thumb base Osteoarthritis (OA). The design will be a prospective longitudinal cohort study linked with a qualitative interview and focus group study. Four NHS sites will recruit 150 people with symptomatic thumb base OA. The primary outcome is the AUSCAN hand pain scale, additionally baseline assessments will be carried out for measures of hand function, quality of life and known musculoskeletal prognostic factors. The study endpoint is six months. Outcome assessments will be conducted by postal/online questionnaire (as applicable) at three and six months. The qualitative and quantitative results from this study will be integrated and presented to a stakeholder group meeting, where participants will be guided to generate recommendations for future care.

Objectives

1. To determine the 6-month outcomes (change in pain, hand function, participation in social roles and activities, and quality of life) in a cohort of patients with thumb base OA receiving supported self-management in specialist NHS services. And to estimate the proportion of those who respond after treatment.
2. To evaluate patient experiences with care and determine what factors patients and clinicians perceive contribute to outcome (candidate prognostic factors).
3. To investigate the association of prognostic factors with pain and function outcomes.
4. To integrate qualitative and quantitative findings to generate recommendations for optimising current care.

STUDY DESIGN

This study is a mixed methods convergent parallel design, and is divided into three parts:

1. Prospective cohort study in people with symptomatic thumb base OA receiving a supported self-management programme to provide 3- and 6-month outcome data; and record any subsequent stepped care provided according to existing guidelines.
2. Qualitative Research: semi-structured interviews will describe the experience of care and explore patient perception of factors related to outcome, and a focus group will explore treating therapist perceptions of factors related to outcome.
3. Stakeholder and PPIE meeting to discuss and disseminate the results with patients and clinicians and to generate recommendations for improving care for patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic thumb base OA, confirmed with at least one of the following clinical signs:

  * Hard tissue enlargement of the thumb carpometacarpal joint
  * Squaring at the base of the thumb
  * Crepitus on movement of the thumb carpometacarpal joint
  * Positive adduction provocation test
  * Positive extension provocation test
  * Positive pressure shear test
  * Pain on palpation of the dorso-radial aspect of the thumb carpometacarpal joint
* Able to give written informed consent.
* Available to attend Occupational Therapy/Physiotherapy/Hand Therapy sessions.

Exclusion Criteria:

* Currently receiving therapy care for thumb base OA.
* Fractures or significant injury or surgery to the wrist or hand on the included side in the previous 6 months.
* Previous surgery to the basal thumb joint on the included side.
* Red flags i.e., diagnosed rheumatic condition (gout, rheumatoid arthritis), progressive neurological signs, any acutely swollen hand joint, serious illness, or disease.
* Participants of any drug or medical device trial in the last 12 weeks.
* Recent steroid injection in their included basal thumb joint (2 months prior to baseline appointment).

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will recruit participants seeking care for a painful thumb, with a clinical diagnosis (signs and symptoms) of thumb base OA. Radiographs are not required to diagnose and provide therapy treatment for thumb base OA, clinical assessment alone will be used (NICE guidelines).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Australian Canadian Osteoarthritis Hand Index (AUSCAN) Hand Pain Subscale | 6 months
  The AUSCAN is a patient-rated, disease-specific, and hand-specific questionnaire with a pain subscale comprising of five items measuring hand pain (0-20), greater scores indicate worse pain.

SECONDARY OUTCOMES:
Osteoarthritis Research Society International (OARSI) responder Criteria | 3 & 6 months
  Participants are evaluated as a responder or non-responder to treatment. This is calculated based on a global rating of change (GROC) question with 6 items (on a Likert scale ranging from completely recovered to much worse); and absolute or relative changes in AUSCAN scores for pain and function (Ref Pham 2004).
Australian Canadian Osteoarthritis Hand Index (AUSCAN) Hand Pain & Function Subscales | 3 & 6 months
  The AUSCAN is a patient-rated, disease-specific, and hand-specific questionnaire comprising of five items measuring hand pain (0-20), one item measuring stiffness (0-4), and nine measuring hand function (0-36). The total score ranges from 0-60 with higher scores indicating more pain, stiffness, or functional limitation.
Numerical rating scale (NRS) Thumb pain (0-10) | 3 & 6 months
  NRS specific to thumb pain severity over the last week, higher scores indicate greater pain severity.
Thumb Pain Frequency | 3 & 6 months
  5 point Likert scale (never- always)
PSEQ | 3 & 6 months
  Pain self efficacy questionnaire
EQ-5D-5L | 3 & 6 months
  Generic health status and quality of life
PROMIS SF | 3 & 6 months
  Social participation and difficulty in daily life

OTHER OUTCOMES:
Prognostic factor analysis | 6 months
  Candidate prognostic factors for response to conservative management will be collected at baseline only. These factors have been identified from a systematic review of the prognosis for pain and function in hand and thumb base OA (61). The prognostic factors fall into the following categories clinical signs, general health, psychological factors, and perceived symptom severity.
The Osteoarthritis Quality Indicator (OA-QI) | 3 & 6 months
  The OA-QI questionnaire will be used to assess patient-perceived quality of care.
Qualitative data | 3-6 months
  Topic guides have been created to explore the expereince of receiving care and on participant and therapist perceived prognostic factors.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Pulvertaft Hand Centre, Derby
  - MOSAIC Service, Nottingham City Care, Nottingham
  - Pennine MSK Partnership Ltd, Oldham
  - Kings Mill Hospital, Hand Therapy Service, Sutton in Ashfield

IPD SHARING:
Plan to Share IPD: Undecided
The data is not being uploaded to an external repository. Keele University have a process for data sharing, and all requests would follow their usual process. The CTU can be contacted from the website https://www.keele.ac.uk/ctu/

REFERENCES:
- See also: 12 NICE Guidelines: osteoarthritis in the over 16s diagnosis and management — https://www.nice.org.uk/guidance/ng226
- See also: TOPS study website for participants — http://thetops.study